CLINICAL TRIAL: NCT00671229
Title: Nitric Oxide, LPS and the Pathogenesis of Asthma Phase 1
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Sandler Program for Asthma Research (Other)
Responsible Party: Marc C. Levesque, NIEHS
Other Study IDs: 12496-CP-006A; Pro00005046
Record Dates: First submitted 2008-05-02; First posted 2008-05-05 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Healthy; Asthma
Keywords: Healthy; Asthma; Nitric Oxide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples, DNA, Exhaled Breah Condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: African American
- 2: Caucasian

SUMMARY:
The purpose of the study is to determine the role of nitric oxide (NO) in asthma. We determine the effect of promoter polymorphisms in the gene for the NO producing enzyme, nitric oxide synthase (NOS2), on exhaled NO in healthy African Americans and Caucasians. We compare exhaled NO levels between African Americans and Caucasians. Information on race or ethnicity, serum samples, blood pressure, exhaled breath condensate and health questionnaires will be collected.

DETAILED DESCRIPTION:
The purpose of the study is to determine the role of nitric oxide (NO) in asthma. We determine the effect of promoter polymorphisms in the gene for the NO producing enzyme, nitric oxide synthase (NOS2), on exhaled NO in healthy African Americans and Caucasians. We compare exhaled NO levels between African Americans and Caucasians. Information on race or ethnicity, serum samples, blood pressure, exhaled breath condensate and health questionnaires will be collected.

Three single nucleotide polymorphisms (SNPs) have been identified in Africans that are associated with increases in systemic NO production. These studies determine whether the NOS2 promoter SNPs are associated with differences in basal exhaled NO levels. The study of exhaled NO levels in individuals with asthma is confounded by the presence of cell types besides bronchial epithelium that produce NO, by differences in the severity of asthma and by the use of medications such as corticosteroids which alter exhaled NO levels.

Therefore, in this study exhaled NO levels in asymptomatic healthy African Americans and Caucasians are measured. The initial analysis of exhaled NO levels indicate that a subset of African American samples contained lower levels of NO than previous measurements of exhaled NO levels in Caucasians. Because differences in exhaled NO levels may influence bronchodilation and other airway responses, as part of this study, the exhaled NO levels of the African American subjects are compared to the results of sample collections from Caucasian samples.

In addition to measures of exhaled NO levels, information on race or ethnicity and DNA samples are collected to characterize samples collected from African American and Caucasian subjects. Serum samples, measures of blood pressure and exhaled breath condensate samples are collected from African Americans and Caucasians to control for confounding variables. Repeated measures of exhaled NO levels are collected to control for fluctuations in exhaled NO levels related to upper respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

* Willing/able to give informed consent
* self declared non-atopic, non-asthmatic
* never cigarette smoker,
* no significant occupational exposure to respiratory irritants or toxins,
* no chronic illness
* no chronic use of medications (excluding contraceptive medication),
* no historical unstable cardiac or severe lung disease,
* within study age parameters of 18 - 40

Exclusion Criteria:

* occupational exposure to hay or grain
* smoked 20 or more packs of cigarettes in a lifetime.
* prior allergen immunotherapy
* Allergy and or asthma
* Students or employees under direct supervision by protocol investigators are ineligible
* Nursing mothers
* pregnancy
* Other investigational medication within the last 30 days
* Other medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2003-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc C Levesque, M.D., PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Levesque MC, Hauswirth DW, Mervin-Blake S, Fernandez CA, Patch KB, Alexander KM, Allgood S, McNair PD, Allen AS, Sundy JS. Determinants of exhaled nitric oxide levels in healthy, nonsmoking African American adults. J Allergy Clin Immunol. 2008 Feb;121(2):396-402.e3. doi: 10.1016/j.jaci.2007.09.031. Epub 2007 Nov 26. PMID 18036642